CLINICAL TRIAL: NCT04453969
Title: Is COVID-19 Transmitted Through Human Milk? Implications for Breastfeeding and Human Milk Banking-Study 1a
Status: Completed | Type: Observational
Sponsor: Deborah O'Connor (Other)
Collaborators: University of Toronto (Other); Sinai Health System (Other)
Responsible Party: Sponsor-Investigator, Deborah O'Connor, Scientist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 39373-a
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV2; Breastmilk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breastfeeding mothers positive for COVID-19
  Interventions: Other: COVID-19

INTERVENTIONS:
Other: COVID-19 — Exposure of interest for this observational study is current COVID-19 positive status or COVID-19 positive status during pregnancy

SUMMARY:
The Canadian Paediatric Society recommends breastfeeding during COVID-19 infection. Human milk is the best form of infant nutrition providing significant protection against many illnesses for term and preterm infants. The impact of a pandemic on breastfeeding is unknown. This study seeks to address this public health issue. Breastmilk will be collected from mothers positive for COVID-19. Samples will be analyzed for the COVID-19 virus specific nucleic acid and antibody in real-time and results will be immediately disseminated to relevant organizations to inform local, national and international guidelines surrounding breastfeeding to protect the health of infants.

ELIGIBILITY:
Inclusion Criteria:

* Current COVID-19 positive status or COVID-19 positive status during pregnancy
* Intent to breastfeed or currently breastfeeding

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-05-24 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Presence of SARS-CoV-2 in breastmilk | 2-6 months
  To describe the presence of SARS-CoV-2 nucleic acid in human milk samples collected from mothers positive for COVID-19
SARS-CoV-2 antibody in breastmilk | 2-6 months
  To describe the presence of SARS-CoV-2 antibody in human milk samples collected from mothers positive for COVID-19

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Sinai Health System, Toronto, Ontario
  - University of Toronto, Toronto, Ontario

REFERENCES:
- [Background] Ismail S, Unger S, Budylowski P, Poutanen S, Yau Y, Jenkins C, Anwer S, Christie-Holmes N, Kiss A, Mazzulli T, Johnstone J, McGeer A, Whittle W, Parvez B, Gray-Owen SD, Stone D, O'Connor DL. SARS-CoV-2 antibodies and their neutralizing capacity against live virus in human milk after COVID-19 infection and vaccination: prospective cohort studies. Am J Clin Nutr. 2024 Feb;119(2):485-495. doi: 10.1016/j.ajcnut.2023.10.008. Epub 2023 Dec 14. PMID 38309831